CLINICAL TRIAL: NCT05015569
Title: A Randomized, Single-Blinded, Continuous Case Series Study to Examine the Impact of Surgical Garment Selection on Patients' Perception of Their Surgical Experience
Brief Title: Compare Patients' Perception of Surgical Experience Based on Garment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: More Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: COVR202011092.3
Record Dates: First submitted 2021-02-02; First posted 2021-08-20 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-08

CONDITIONS: Anxiety; Orthopedic Disorder
Keywords: anxiety; modesty; dignity; satisfaction
MeSH Terms: conditions — Anxiety Disorders; Musculoskeletal Diseases; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Treatment allocation will be determined using a block randomized crossover trial design.
Who Masked: Participant
Masking Description: Patients will be blinded to the difference between garment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Patient Gown + COVR garment (Active Comparator): Patients will receive the standard of care patient gown and a COVR garment. Patients undergoing unilateral lower extremity surgery will receive a half short. Patients undergoing upper extremity or spine surgery will receive the brief (bilateral) style COVR garment.
  Interventions: Device: COVR Medical Garment; Other: Standard Patient Gown
- Patient Gown (Active Comparator): Patient will receive the standard of care patient gown only without undergarments.
  Interventions: Other: Standard Patient Gown

INTERVENTIONS:
Device: COVR Medical Garment — COVR undergarments are available in a "Half Short" design for unilateral lower extremity procedures and a "Bilateral" (brief) style garment designed for bilateral lower extremity procedures. Either style may be worn for upper extremity, trunk, spine procedures, etc. where an undergarment would be preferred along with a standard hospital gown. The garments are available in a variety of sizes. The COVR garments can be released at the hip(s)/waistline for improved access to the lateral hip and include retractable panels for procedural access to the groin and genitals if needed by the care team.
  Arms: Patient Gown + COVR garment
Other: Standard Patient Gown — The standard patient gown is provided to all patients in a hospital setting.

SUMMARY:
This study seeks to compare how patients rank perception of anxiety, modesty, dignity and overall satisfaction when patients are provided with either a standard patient gown or a standard patient gown plus a pair of specialized surgical undergarments (COVR Medical) for orthopedic surgical procedures.

DETAILED DESCRIPTION:
Given the movement in patient modesty, and the limited number of studies focused specifically on how preserving patient modesty/privacy impacts the patient's perception of the hospital experience, targeted studies with larger sample sizes are clearly needed to better understand these complex interactions. This study seeks to compare how patients rank perception of anxiety, modesty, dignity and overall satisfaction when patients are provided with either a standard patient gown or a standard patient gown plus specialized surgical undergarments (COVR Medical) for orthopedic surgical procedures. The investigators hypothesize that the group with the standard patient gown plus a specialized surgical undergarment will have lower anxiety and increased perception of modesty, dignity, and satisfaction. A secondary objective is to determine whether there is a difference in treatment surgical subgroups regarding anxiety, modesty, dignity, and overall satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo surgery by a musculoskeletal surgeon at The CORE Institute orthopedic Specialty Hospital (CISH).
* Adults 18 years or older.
* Will receive orthopedic surgery of the lower extremity, upper extremity or spine.
* Speaks, reads, and understands English
* Enrolled pre-operatively within 3 weeks of surgery date.

Exclusion Criteria:

* Unwilling to provide informed consent.
* Unwilling to participate in surveys.
* Body habitus outside of the COVR medical size range. (See Appendix 1)
* Procedure that does not meet the medical billing and coding definition of Surgery.
* Incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall perception of anxiety, modesty, privacy, and satisfaction | Within 2 hours before surgery
  7 question surveys designed for this study
Overall perception of anxiety, modesty, privacy, and satisfaction | Up to 1 week
  7 question surveys designed for this study

CONTACTS AND LOCATIONS:
Overall Officials: Marc Jacofsky, PhD, Principal Investigator — More Foundation
Locations (1):
- The CORE Institute, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared.